CLINICAL TRIAL: NCT03931356
Title: Follow-up of Pulmonary Toxicity by Respiratory Functional Tests of Patients Treated With Dynamic Cancer ARCtherapy for Bronchopulmonary Cancer.
Brief Title: Follow-up of Pulmonary Radiotoxicity for Bronchopulmonary Cancer.
Acronym: TEFRARC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29 BRC17.0167
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cancer, Lung; Radiotherapy; Complications
MeSH Terms: conditions — Lung Neoplasms | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pulmonary function tests — analysis of lung volume and diffusion capacity

SUMMARY:
assess the consequences of low doses of radiation delivered by the volumetric radiotherapy, on the respiratory capacity of patients treated for bronchopulmonary carcinoma, by a follow up of functional respiratory exploration.

DETAILED DESCRIPTION:
Radiation therapy with or without chemotherapy is a stable treatment in the management of patients with localized smack cell bronchopulmonary cancers, or not to small cells not metastatic but not operable. Radiation therapy results in changes in respiratory function, as measured by respiratory function tests and represented primarily by spirometry, total body plethysmography, and the diffusion capacity of the alveolar-capillary membrane.

Although these tests are minimally invasive, few studies have investigated the implications of radiation therapy on lung function in patients treated for pulmonary neoplasia, while these patients are often already carriers of respiratory diseases and will receive further chemotherapy during their illness, subject to their general good condition, including respiratory. No method has been recognized as superior for measuring the consequences of radiation therapy on respiratory function. After chest radiotherapy alone, the decline in diffusion capacity is estimated at 10-34%. New irradiation techniques have emerged over the last decade, in particular dynamic arc therapy. This innovative technology, combined with image-guided irradiation processes, ensures high-precision, short-term treatment, but exposes virtually all of the lungs to irradiation, although at very low doses, the objective consequences of which on respiratory functional explorations have never been reported.

The aim of this study is therefore to assess the consequences of low doses of radiation delivered by this recent technology, volumetric therapy, on the respiratory capacity of patients treated with radiotherapy within the framework of of bronchopulmonary carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* bronchopulmonary carcinoma histological proved
* OMS 0-2
* indication of radio(chimio)therapy alone approved by multidisciplinary comitee
* non opposition formular completed

Exclusion Criteria:

* SBRT indication
* history of thoracic surgery or irradiation
* unstable disease
* oxygenotherapy dependance
* severe chronic bronchitis
* collagen disease
* pregnancy
* contraception refusal
* refusal or incapacity to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with bronchopulmonary carcinoma treated by radio(chimio)therapy alone
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
diffusion capacity | 3 months
  diminution of 20% or more of the diffusion capacity at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest (Morvan), Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement